CLINICAL TRIAL: NCT01317706
Title: Comparison Between Ultrasonographic Cervical Length and Bishop Score in Preinduction Cervical Assessment
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Seoul National University Bundang Hospital, Department of Obstetrics and Gynecology, Seoul National University Bundang Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Diagnostic
Other Study IDs: BS_CL_01
Record Dates: First submitted 2011-03-16; First posted 2011-03-17 (Estimated); Last update posted 2011-03-17 (Estimated); Status verified 2011-03

CONDITIONS: Failed Induction of Labor
Keywords: Bishop score, Cervical length, Cervical ripening, Labor induction

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No

ARMS (2):
- Bishop score (Active Comparator)
  Interventions: Other: Assessment of cervical status
- transvaginal ultrasound (Active Comparator)
  Interventions: Other: Assessment of cervical status

INTERVENTIONS:
Other: Assessment of cervical status — Assessment of cervical status based on Bishop score versus sonographically measured cervical length

SUMMARY:
To compare the ultrasonographic cervical length with the Bishop score in determining the administration of prostaglandin for preinduction cervical ripening in nulliparas at term.

ELIGIBILITY:
Inclusion Criteria:

* nulliparous patients
* singleton pregnancy
* live fetus with vertex presentation
* intact amniotic membranes
* > 37 weeks gestation
* absence of labor
* no previous uterine surgical procedures

Exclusion Criteria:

* major congenital anomaly

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 154 (Actual)
Dates: Start 2008-11; Primary Completion 2010-08 (Actual); Study Completion 2010-08 (Actual)

PRIMARY OUTCOMES:
Successful labor induction | Eleven hours of initiating oxytocin on the fist day of induction
  Induction success was defined as an ability to achieve the active phase of labor corresponding to a cervical dilatation of ≥ 4 cm within 11 hours of initiating oxytocin (i.e., within 22 hours of the administration of a dinoprostone vaginal insert) on the first day of induction.

SECONDARY OUTCOMES:
the need for oxytocin induction | After removing prostaglandin, the following day when an intravenous oxytocin infusion was started
  1. the interval from start of oxytocin to the active phase of labor
  2. the interval from start of oxytocin to delivery
  3. vaginal delivery within 24 hours of starting induction
  4. the incidence of cesarean delivery

CONTACTS AND LOCATIONS:
Overall Officials: Kyo Hoon Park, MD, PhD, Principal Investigator — Seoul National University Bundang Hospital
Locations (1):
- Department of Obstetrics and Gynecology Seoul National University Bundang Hospital, Seongnam-si, Gyeonggi-do, South Korea